CLINICAL TRIAL: NCT04254731
Title: The Study of Potential Normalization of Cardiac Rhythm Following Drug Exchange From Chimeric Methadone to Active Methadone
Brief Title: Effects of Switching From Racemic Methadone to R-methadone on QTc Intervals
Acronym: MePhaCard
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mimi Stokke Opdal, Senior Consultant and Associate Professor of Clinical Pharmacology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/793 REK
Record Dates: First submitted 2020-01-06; First posted 2020-02-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Adverse Drug Effect; Drug Effect; Heart Arrhythmia
Keywords: Racemic methadone; R-methadone; QTc interval; Methadone maintenance treatment patients
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Arrhythmias, Cardiac | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Patients included were stabilized on per os methadone maintenance treatment and had automatically ECG recorded QTc interval greater or equal to 450 ms. The patients were switched to pure R-methadone per os (half dose of the racemic methadone used). Doses, serum drug concentrations, QTc-time were recorded before and after drug switch. Serum-electrolytes (Mg, K, Ca) and opioid withdrawal symptom scale (OWS) were also measured and scored before and after drug switch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cross over study before and after drug switch (Other): Stabilized on racemic methadone dose, switched to R-methadone of half racemic methadone dose. Cross over study, own control
  Interventions: Drug: Same individuals treated with racemic methadone and switched to levomethadone (R-methadone)

INTERVENTIONS:
Drug: Same individuals treated with racemic methadone and switched to levomethadone (R-methadone)
  Other Names: Drugs provided from the pharmaceutical company called DnePharma AS (Den norske Eterfabrikk ( DnE), address Karihaugen 22, Oslo, Norway, drug delivered to patient from home nurse or pharmacy

SUMMARY:
Effects of switching from racemic methadone to R-methadone on serum methadone concentrations and QTc intervals

DETAILED DESCRIPTION:
Racemic methadone may prolong the QTc interval, which is associated with fatal arrhythmias. In vitro studies have shown that R-methadone has less inhibitory effect than S-methadone on the voltage-gated potassium channel current, and is thus thought to have less effect on the QTc interval.

The investigators hypothesized that switching from racemic to R-methadone would reduce the methadone serum concentration and also its effect on the QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* Stabilized on daily methadone dose
* Not using other drugs of abuse
* QTc-time recorded automatically, patient inclusion if QTc interval was greater or equal to 450 ms
* Older than 18 years
* Can sign and understand a written Consent

Exclusion Criteria:

* Can not cooperate regarding observed daily drug intake
* Serious psychiatric disease
* Untreated serious somatic disease
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Effects of switching from racemic methadone to R-methadone on serum methadone concentrations. | Time frame of each patient form inclusion to end study was 35-40 days.
  Ten patients stabilized on racemic methadone dose were switched to R-methadone and effects on serum methadone concentrations were studied. Methadone concentrations (nmol/L) were measured by validated high pressure liquid chromatography coupled to mass spectrometry detection (LC-MSMS).
Effects of switching from racemic methadone to R-methadone on QTc interval | Time frame of each patient form inclusion to end study was 35-40 days.
  In ten patients QTc intervals were recorded on racemic methadone treatment at Cmin and Cmax of methadone drug concentrations and likewise after the shift to R-methadone. QT intervals (ms) on ECG were recorded automatically and read manually by experienced cardiologists.
Effects of switching from racemic methadone to R-methadone on opioid withdrawal symptoms (OWS) | Time frame of each patient form inclusion to end study was 35-40 days.
  Ten patients: each patients had OWS recorded on racemic and R-methadone treatment using OWS.
Effects of switching from racemic methadone to R-methadone, stability of serum electrolytes (Ca, Mg, K) in patients | Time frame of each patient form inclusion to end study was 35-40 days.
  Ten patients: samples for serum electrolytes were collected before and after switch to R-methadone. Measured by routine analysis at Cobas 8000 (unit mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Stokke S Opdal, MD, PhD, Study Director — Oslo University Hospital and University of Oslo; Peter Krajci, MD, PhD, Study Director — Oslo University Hospital
Locations (3):
- Norway (3):
  - Department of Pharmacology , Oslo University Hospital, Oslo
  - Department of Pharmacology and Department of Substance Use Disorder, Oslo University Hospital, Oslo
  - Department of Substance Use Disorder, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared when the manuscript has been accepted for publication.
Supporting Information: Study Protocol
Time Frame: Protocol in Norwegian attached
Access Criteria: IPD proving the results of the different outcome measures will be shared, see above

REFERENCES:
- [Background] Havig SM, Berg-Pedersen RM, Krabseth HM, Muller LD, Haugaa K, Zare HK, Gjesdal K, Krajci P, Opdal MS. Effect on QTc interval by switching from methadone to equipotent R-methadone dose in methadone maintenance treatment patients. Basic Clin Pharmacol Toxicol. 2024 Apr;134(4):519-530. doi: 10.1111/bcpt.13982. Epub 2024 Feb 3. PMID 38308508
- See also: abstract from EACPT 2019, see abstract 1168 — https://link.springer.com/content/pdf/10.1007%2Fs00228-019-02685-2.pdf

DOCUMENTS (2):
  • Study Protocol (2012-04-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04254731/Prot_000.pdf
  • Informed Consent Form (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT04254731/ICF_001.pdf